CLINICAL TRIAL: NCT05963503
Title: Investigation of Relationship Between Health Literacy and Physical Activity, Anxiety and Depression, Adherence to Airway Clearance Techniques in Adult Patients With Cystic Fibrosis
Brief Title: Relationship Between Health Literacy and Physical Activity in Adult Patients With Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aydan Aslı Aksel Uylar, Physiotherapist, Hacettepe University
Other Study IDs: GO 22/114
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Inclusion Criteria:
  have a confirmed diagnosis of CF stable clinical condition 18-65 ages volunteering to participate
  Exclusion Criteria:
  having a serious comorbidity that limits mobilization or participation in physical activity being illiterate having cognitive problems being pregnant incomplete answers to surveys
  Interventions: Other: Assessments
- Controls: Inclusion Criteria:
  18-65 ages volunteering to participate
  Exclusion Criteria:
  having any cardiopulmonary disease having cognitive problems being illiterate
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — Health literacy Anxiety and depression Physical activity Adherence to airway clearance techniques

SUMMARY:
The purpose of this study investigation of relationship between health literacy and physical activity, anxiety and depression, adherence to airway clearance techniques in adult patients with cystic fibrosis.

DETAILED DESCRIPTION:
The assessment will begin with demographic information then health literacy, depression and anxiety and physical activity level will evaluation with related questionnaires.

ELIGIBILITY:
Inclusion Criteria:

be between the ages of 18-65 volunteering to participate

Exclusion Criteria:

having any cardiopulmonary disease having cognitive problems being illiterate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cystic fibrosis and healthy participants between 18-65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Health Literacy | 5 minutes
  Health literacy will be evaluated with Health Literacy Scale. This scale total score ranges from 25-125 and lower scores show that lower health literacy.

SECONDARY OUTCOMES:
Anxiety and Depression | 5 minutes
  Anxiety and depression will be evaluated with Hospital Anxiety and Depression Scale. A score of 11 or more indicates mood disorders. Anxiety or depression subscales score ranges from 0-21.
Physical Activity | 3 minutes
  Physical activity will be evaluated with International Physical Activity Questionnaire Short Form.
Adherence to Airway Clearance Tecniques | 1 minute
  Frequency of used airway clearance tecniques for a week

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar Yağlı, Study Director — Hacettepe University; Ebru Damadoğlu, Study Chair — Hacettepe University; Oğuz Karcıoğlu, Study Chair — Hacettepe University; Aydan Aslı Aksel Uylar, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)